CLINICAL TRIAL: NCT05420324
Title: A Multicenter, Single-arm, Open-label Phase II Study to Evaluate the Efficacy and Safety of YH003 in Combination with Pebolizumab and Albumin Paclitaxel in First-line Treatment of Patients with Unresectable/metastatic Mucosal Melanoma
Brief Title: A Study to Assess YH003 in Combination with Pebolizumab and Albumin Paclitaxel Injection in Subjects with Unresectable/metastatic Mucosal Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eucure (Beijing) Biopharma Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: YH003006
Record Dates: First submitted 2022-06-07; First posted 2022-06-15 (Actual); Last update posted 2025-01-06 (Actual); Status verified 2025-01

CONDITIONS: Mucosal Melanoma
MeSH Terms: interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intervention/treatment (Experimental): YH003 in combination with pebolizumab and albumin paclitaxel in first-line treatment of patients with unresectable/metastatic mucosal melanoma
  Interventions: Drug: YH003; Drug: Pembrolizumab; Drug: albumin paclitaxel

INTERVENTIONS:
Drug: YH003 — YH003 will be administered intravenously over 30 minutes every 21-day cycle.
Drug: Pembrolizumab — Pembrolizumab will be administered intravenously over 30 minutes every 21-day cycle.
Drug: albumin paclitaxel — Albumin paclitaxel will be administered intravenously over 30 minutes every 21-day cycle.

SUMMARY:
This study is a multicenter, single-arm, open-label phase II study to assess the efficacy and safety of YH003 in combination with pembrolizumab and nab-paclitaxel in the first-line treatment of patients with unresectable/metastatic mucosal melanoma.

ELIGIBILITY:
Inclusion Criteria:

* 1.Subjects must have the ability to understand and willingness to sign a written informed consent document.
* 2. Subjects must have histologically advanced or cytologically confirmed metastatic or unresectable mucosal melanoma;
* 3.Subjects have not received standard systemic therapy; patients have disease progression 6 months or more after the end of neoadjuvant or adjuvant therapy (except nab-paclitaxel), and can be enrolled in the clinical study;
* 4. Subject must have at least 1 unidimensional measurable disease by RECIST 1.1;
* 5. Subjects must be age 18 years or older;
* 6. Subjects must have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* 7. Life expectancy ≥3 months based on investigator's judgement；
* 8. Subjects must have adequate organ function;
* 9. Women of childbearing potential need to have a negative pregnancy test and need to take contraceptive/contraceptive measures including their partners.

Exclusion Criteria:

* 1.Subjects have another active invasive malignancy within 5 years；
* 2.The subject has received anti-tumor therapy or other investigational drug therapy or traditional Chinese medicine (herbal medicine) with anti-tumor indications prior to the first dose;
* 3.Subjects with a history of ≥ Grade 3 immune-related adverse events resulted from previous immunotherapy.
* 4.History of clinically significant sensitivity or allergy ；
* 5.Primary central nervous system (CNS) malignancies or symptomatic CNS metastases.；
* 6.History of (non-infectious) pneumonitis that required corticosteroids or current pneumonitis, or history of interstitial lung disease；
* 7.Subjects have active pulmonary embolism with hemodynamic changes 12 weeks before the first dose;
* 8. Subjects must not have a known or suspected history of autoimmune disease within 3 years prior to the first dose of study treatment;
* 9. Subjects have clinically uncontrolled diseases;
* 10. Subjects have severe cardiovascular disease;
* 11. Subjects have evidence of active infection;
* 12. Subjects must not have a known or suspected history of an autoimmune disorder；
* 13.Major surgery within 4 weeks prior to study entry and Minor surgery within 2 weeks prior to the first dose.
* 14. Any condition that the investigator assesses as inappropriate for participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-06-13 (Actual); Primary Completion 2024-03-04 (Actual); Study Completion 2024-03-04 (Actual)

PRIMARY OUTCOMES:
Confirmed Objective Response Rate (ORR) | up to 2 years
  Overall Response Rate (ORR) by investigator's assessment according to the Response Evaluation Criteria in Solid Tumors (RECIST) v1.1

CONTACTS AND LOCATIONS:
Locations (12):
- China (12):
  - Cancer Hospital of Fujian, Fuzhou, Fujian
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - Cancer Hospital of Zhenzhou, Zhengzhou, Henan
  - Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Hunan Cancer Hospital, Changsha, Hunan
  - The First Hospital of Jilin University, Jilin, Jilin
  - The First affiliated Hospital of Dalian Medical University, Dalian, Liaoning
  - Nanjing Drum Tower Hospital, Nanjing, Nanjing
  - West China Hospital of Sichuan University, Chengdu, Sichuan
  - Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality
  - Yunnan Cancer Hospital, Kunming, Yunnan
  - Cancer Hospital of The University of Chinese Academy of Sciences, Hangzhou, zhenjiang

IPD SHARING:
Plan to Share IPD: No